CLINICAL TRIAL: NCT00829478
Title: Improving Quality of Care for Atrial Fibrillation by Promoting Patient-Centered Decision Making
Brief Title: Improving the Quality of Care for Atrial Fibrillation by Promoting Patient-Centered Decision Making
Acronym: AFIB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: Donaghue Medical Research Foundation (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Fried0011
Record Dates: First submitted 2009-01-24; First posted 2009-01-27 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cerebrovascular accident; Anticoagulation; Decision-making
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Usual Care
  Interventions: Other: Usual Care
- 2 (Experimental): Intervention
  Interventions: Behavioral: Decision Aid for Atrial Fibrillation

INTERVENTIONS:
Behavioral: Decision Aid for Atrial Fibrillation — Single contact educational session
  Arms: 2
Other: Usual Care — Usual Care
  Arms: 1

SUMMARY:
The primary aim of this proposal is to determine the effectiveness of a decision support tool on improving the process of shared decision-making for treatment on nonvalvular atrial fibrillation (NVAF) compared to receipt of usual care.

DETAILED DESCRIPTION:
Decision-making regarding appropriate therapy for non-valvular atrial fibrillation (NVAF) is a complex process. Different options carry with them different profiles of risks and benefits, and choosing the "right" therapy depends upon the patient's understanding of these risks and benefits and a consideration of the risks and benefits according to the patient's values and preferences. Studies have shown that patients' preferred therapy frequently disagrees with what is recommended by disease management guidelines.

The purpose of this study is to examine an intervention to improve the quality of decision-making for NVAF compared to usual care. The intervention has several components, including: a) educating the patient about why values and preferences are important to the decision-making process, b) providing an individualized assessment of the risks and benefits of each of the treatment options, c) exploring patients' values and preferences as they relate to the risks and benefits of each of the treatment options, d) preparing the patient to discuss his/her preferences with the physician.

ELIGIBILITY:
Inclusion Criteria:

* 45 years or older
* Be scheduled to see primary Doctor at VA
* Diagnosis of atrial fibrillation
* English speaking

Exclusion Criteria:

* Have valvular disease as the cause of Afib
* Be on warfarin for a condition other than NVAF
* Have a contraindication to warfin
* Have a contraindication to ASA
* Life expectancy of less than 12 months
* Cognitive impairment
* Receiving anti-platelet agent other than aspirin
* Receiving care in a supervised resident clinic or from an attending physician who refuses participation in the study
* Bleed with identified source in the last 12 months
* Bleed with an unidentified source
* History of intracerebral hemorrhage
* Severe hearing impairment
* Severe visual impairment

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | Immediately following and 1-month post-intervention

SECONDARY OUTCOMES:
Knowledge regarding atrial fibrillation | Immediately following study intervention and 1 month post-intervention
Anxiety | Immediately following intervention and 1 month post-intervention
Changes in treatment plan for atrial fibrillation | Within 30 days post-intervention
Quality of clinician-patient communication | Clinician visit immediately post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Terri R Fried, M.D., Principal Investigator — VA Connecticut HS
Locations (1):
- VA Connecticut Healthcare System - West Haven Campus, West Haven, Connecticut, United States